CLINICAL TRIAL: NCT06982053
Title: [68Ga]Ga-GZP PET and [18F]FDG PET for Early Response Prediction in Locally Advanced Rectal Cancer Undergoing Neoadjuvant Short-Course Radiotherapy Plus Immunochemotherapy: A Single-center Clinical Study
Brief Title: [68Ga]Ga-GZP PET for Early Response Prediction in Colorectal Cancer During Neoadjuvant Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0506
Record Dates: First submitted 2025-05-09; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer Control and Prevention; Colorectal Cancer Recurrent; Colorectal Cancer Metastatic; Colorectal Cancer Screening
Keywords: Neoadjuvant therapy; Immunotherapy; PET; PET/CT; PET/MR; Granzyme B; Colorectal cancer; Locally advanced rectal cancer
MeSH Terms: conditions — Lipodystrophy, Congenital Generalized; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Received 68Ga-NOTA-GZP PET scanning (Experimental)
  Interventions: Diagnostic Test: Received 68Ga-NOTA-GZP PET scanning

INTERVENTIONS:
Diagnostic Test: Received 68Ga-NOTA-GZP PET scanning — Received twice 68Ga-NOTA-GZP PET scanning before neoadjuvant therapy and radical surgery.
  Other Names: Received 18F-FDG PET scanning

SUMMARY:
This diagnostic study investigates the value of 68Ga-NOTA-GZP PET imaging in predicting and evaluating immunotherapy response in malignant tumors by enrolling pathologically confirmed patients scheduled for immunotherapy and healthy volunteers. All participants underwent immunohistochemical staining of tumor tissue for immune checkpoint markers (PD-1 or CTLA-4) and granzyme B expression prior to signing informed consent for 68Ga-NOTA-GZP PET imaging. Patients received baseline scans before initial immunotherapy and follow-up scans during treatment cycles 2-4, with clinical monitoring continuing until 6 months post-treatment, while healthy volunteers completed single scans with pharmacokinetic analysis through serial blood/urine sampling. Comprehensive data collection included demographic information, clinical characteristics, immunohistochemistry results, laboratory tests (blood routine, liver/kidney function), PET imaging findings, and other relevant imaging data, with treatment response ultimately assessed according to RECIST 1.1 and iRECIST criteria at the 6-month follow-up endpoint.

DETAILED DESCRIPTION:
Malignant tumors represent one of the leading causes of mortality worldwide, posing a significant threat to human health, where early diagnosis and timely intervention can substantially improve clinical outcomes. In recent years, immunotherapy has emerged as a cornerstone in comprehensive cancer treatment, with immune checkpoint inhibitors (ICIs) serving as a primary therapeutic modality. ICIs function by targeting regulatory pathways of T cells, specifically through blockade of immune checkpoints to enhance cytotoxic T cell activity and thereby elicit anti-tumor immune responses. However, the clinical benefits remain limited to a subset of patients, with many eventually experiencing disease progression or recurrence. Given the heterogeneous response patterns observed during immunotherapy, early and dynamic treatment response assessment becomes paramount - early identification of responders versus non-responders enables timely stratification of patients to avoid ineffective treatments, while continuous monitoring allows for comprehensive evaluation of tumor response patterns to minimize unnecessary adverse effects.

The cytotoxic lymphocytes play a pivotal role in anti-tumor immunity, with granzyme B, a serine protease released by activated cytotoxic lymphocytes during immune responses, representing one of the two principal mechanisms through which lymphocytes mediate cancer cell apoptosis. The quantification of granzyme B directly reflects the activity status of cytotoxic lymphocytes. Compared to general immune cell infiltration assessments, measuring active immune cell populations provides a more precise indicator of immune response intensity and greater predictive value for immunotherapy outcomes. The development of 68Ga-NOTA-GZP, a 68Ga-labeled peptide specifically targeting granzyme B, enables non-invasive visualization of cytotoxic lymphocyte activity. This novel PET tracer shows potential for early differentiation between treatment responders and non-responders, facilitating prompt clinical decision-making to discontinue ineffective therapies.

Building upon the promising potential of 68Ga-NOTA-GZP in immunotherapy monitoring, this study aims to systematically evaluate its efficacy in predicting and assessing treatment responses in malignant tumors. Using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) and immune-modified RECIST (iRECIST) as reference standards, we will investigate the tracer's capability for early treatment response prediction and real-time monitoring, with the ultimate goals of accurately stratifying patients at the earliest timepoint and minimizing unnecessary immunotherapy-related toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed treatment-naïve locally advanced rectal adenocarcinoma (T3-4N0M0 or T1-4N+M0)
* No severe hematologic, cardiac, pulmonary, hepatic, or renal dysfunction
* No immunodeficiency diseases
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1

Exclusion Criteria:

* Prior anti-PD-1/PD-L1 antibody therapy
* History of pelvic radiotherapy
* Active autoimmune disease (excluding vitiligo and type 1 diabetes)
* Hypersensitivity to monoclonal antibodies
* History of interstitial lung disease
* Active uncontrolled infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical response | 4 - 6 months.
  Proportion of participants achieving clinical complete response, defined as the absence of detectable tumor residues in both primary lesions and regional lymph nodes through standardized post-neoadjuvant diagnostic evaluations including:
  Endoscopic ultrasound (EUS) Pelvic MRI (T2-weighted imaging with diffusion-weighted sequences) Chest/abdominal CT (RECIST 1.1 criteria)
Pathological response | 4 - 6 months.
  Pathological complete response (pCR) rate determined by histopathological examination
  * ypT0 (no viable tumor cells in primary tumor specimen)
  * ypN0 (no tumor cells in regional lymph nodes) Mandatory whole-mount sectioning of surgical specimens according to CAP (College of American Pathologists) protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan 430022, Hubei Province, China., Wuhan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in primary and secondary outcomes of the study, including:
  * Baseline demographics (age, sex, race)
  * Clinical characteristics (tumor stage, biomarker status)
  * Efficacy outcomes (response rates, progression-free survival)
  * Safety data (adverse events, laboratory parameters)
  * Associated documents
  * PET parameters
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available starting 01/01/2025 with no end date, contingent on repository maintenance and ethical approvals.
Access Criteria: 1. Who can access the data?
  De-identified IPD and supporting documents will be available to researchers with a valid scientific question, provided they:
  * Submit a methodologically sound proposal (with analysis plan)
  * Provide proof of ethics approval from their institution
  * Sign a Data Use Agreement prohibiting re-identification
    2. What data will be shared?
  * Included: Baseline demographics, outcome measures, safety data, study protocol, and data dictionary
  * Excluded: Direct identifiers (names, addresses), raw genomic data
    3. How to access?
    1. Submit request via email
    2. Independent Review Panel evaluates proposals (4-week review period)
    3. Approved users receive de-identified data in CSV/SAS format
    4. Restrictions
  * Prohibited: Commercial use, patient re-identification
  * Required: Citation of original study in publications